CLINICAL TRIAL: NCT06235775
Title: Twelve-months Extension Study to Explore the Long-Term Safety and Efficacy of Subcutaneous Administration of GV1001 1.12 mg/Day in Patients With Progressive Supranuclear Palsy Who Completed Study GV1001-PSP-CL2-011
Brief Title: Administration of GV1001 for the Treatment of Progressive Supranuclear Palsy Who Completed Study GV1001-PSP-CL2-011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV1001-PSP-CL2-011-E
Record Dates: First submitted 2023-12-11; First posted 2024-02-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy GV1001
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GV1001 1.12 mg (Experimental): In GV1001-PSP-CL2-011 study, subjects who were in the trial group (Study Group 1(GV1001 0.56 mg/day), Study Group 2(GV1001 1.12 mg/day) is alternately administered High-dose test drug(GV1001 1.12 mg/day) and placebo once a week from Ex-Visit 1(Visit 16, Week 26) to Ex-Visit 5(Visit 20, Week 30) and High-dose test drugs(GV1001 1.12 mg/day) are administered from Ex-Visit 6 (Visit 21, Week 32) to Ex-Visit 26(Visit 41, Week 72) every two weeks.
  In the GV1001-PSP-CL2-011 study, subjects who were in the placebo group are administered placebo at Ex-Visit 1 (Visit16, Week26), the first visit of the extension study, and Ex-Visit 2 (Visit17, Week27) to Ex-Visit 5 (Visit 20, Week 30), High-dose test drugs(GV1001 1.12 mg/day) are administered once a week and High-dose test drugs (GV1001 1.12 mg/day) are administered from Ex-Visit 6 (Visit 21, Week 32) to Ex-Visit 26(Visit 41, Week 72) every two weeks.
  Interventions: Drug: GV1001 Placebo; Drug: GV1001 1.12mg

INTERVENTIONS:
Drug: GV1001 Placebo — 0.9% normal saline
  Other Names: Normal saline
Drug: GV1001 1.12mg — Lyophilized peptide from hTERT
  Other Names: Tertomotide 1.68mg

SUMMARY:
The study will be conducted by the Sponsor to evaluate Twelve-months Long-Term Safety and Efficacy of GV1001 (1.12 mg) administered subcutaneously as a treatment for Progressive Supranuclear Palsy(PSP). In 75 patients diagnosed with PSP Richardson(PSP-RS) or PSP-Parkinsonism (PSP-P) who Completed Study GV1001-PSP-CL2-011.

DETAILED DESCRIPTION:
In GV1001-PSP-CL2-011 study, subjects who were in the trial group (Study Group 1(GV1001 0.56 mg/day), Study Group 2(GV1001 1.12 mg/day) is alternately administered High-dose test drug(GV1001 1.12 mg/day) and placebo once a week from Ex-Visit 1(Visit 16, Week 26) to Ex-Visit 5(Visit 20, Week 30) and High-dose test drugs(GV1001 1.12 mg/day) are administered from Ex-Visit 6 (Visit 21, Week 32) to Ex-Visit 26(Visit 41, Week 72) every two weeks.

In the GV1001-PSP-CL2-011 study, subjects who were in the placebo group are administered placebo at Ex-Visit 1 (Visit16, Week26), the first visit of the extension study, and Ex-Visit 2 (Visit17, Week27) to Ex-Visit 5 (Visit 20, Week 30), High-dose test drugs(GV1001 1.12 mg/day) are administered once a week and High-dose test drugs (GV1001 1.12 mg/day) are administered from Ex-Visit 6 (Visit 21, Week 32) to Ex-Visit 26(Visit 41, Week 72) every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* A person who has been registered in the GV1001-PSP-CL2-011 clinical trial and has completed administration by Week 24
* A patient who accompanied all visits with the subject for the scheduled visit of this clinical trial, has a guardian who can supervise the subject's compliance with the examination and examination procedures conducted at the time of the visit, and provides information on the subject's indications, and whose guardian has agreed in writing to participate in the clinical trial (except where it is unnecessary to accompany the guardian at the discretion of the investigator)
* Patient and/or representative of the patient who has voluntarily agreed in writing to participate in this clinical trial

Exclusion Criteria:

* Patients deemed unsuitable by the investigator to participate in this extension study
* Pregnant or male subjects who do not consent to contraception by medically approved methods (surgical infertility, intrauterine contraceptive devices, fallopian tube ligature, double blocking (combined use of male condoms, female condoms, cervical caps, contraceptive diaphragm and sponges) and 90 days after clinical trial participation However, women who have undergone menopause or surgical infertility procedures (such as vasectomy and difficult conception on both sides) before participating in clinical trials can participate without consent to contraception.
* Pregnant women or breastfeeding women

Ages: 41 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 12 months
  Adverse Event
Change in Hematological tests WBC(10^3/µl) | 12 months
  WBC(10^3/µl)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests RBC(10^6/µl) | 12 months
  RBC(10^6/µl)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests Hemoglobin(g/dL) | 12 months
  Hemoglobin(g/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests Hematocrit(%) | 12 months
  Hematocrit(%)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests Platelets count(10^3/µl) | 12 months
  Platelets count(10^3/µl)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests WBC differential count (Neutrophils(%)) | 12 months
  WBC differential count (Neutrophils(%)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests WBC differential count( Lymphocytes(%)) | 12 months
  Lymphocytes(%)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests WBC differential count( Monocytes(%)) | 12 months
  Monocytes(%)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests WBC differential count(Eosinophils(%)) | 12 months
  Eosinophils(%)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematological tests WBC differential count(Basophils(%)) | 12 months
  Basophils(%)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests BUN(mg/dL) | 12 months
  BUN(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Creatinine(mg/dL) | 12 months
  Creatinine(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Uric acid(mg/dL) | 12 months
  Uric acid(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Total bilirubin(mg/dL) | 12 months
  Total bilirubin(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Albumin(g/dL) | 12 months
  Albumin(g/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Total Protein(g/dL) | 12 months
  Total Protein(g/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests ALT(U/L) | 12 months
  ALT(U/L)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests AST(U/L) | 12 months
  AST(U/L)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests γ-GTP(U/L) | 12 months
  γ-GTP(U/L)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Alkaline phosphatase(U/L) | 12 months
  Alkaline phosphatase(U/L)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Glucose(mg/dL) | 12 months
  Glucose(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in Hematochemical tests Total Cholesterol(mg/dL) | 12 months
  Total Cholesterol(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in urine tests Protein-Albumin(mg/dL) | 12 months
  Protein-Albumin(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in urine tests Glucose(mg/dL) | 12 months
  Glucose(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in urine tests Ketones(mg/dL) | 12 months
  Ketones(mg/dL)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in urine tests WBC(HPF) | 12 months
  WBC(HPF)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Change in urine tests Blood-RBC(HPF) | 12 months
  Blood-RBC(HPF)
  For the laboratory test results, continuous variables will present the test values at each visit as well as descriptive statistics (number of subjects observed, mean, standard deviation, median, minimum, and maximum) for changes from the baseline(Ex-Visit 1(Visit 16, Week 26) by both integration and treatment group in the extension study. For categorical variables, shift tables will be presented by treatment group
Blood Pressure (mmHG) | 12 months
  Change in Blood Pressure (mmHG)
Pulse rate(beats per min) | 12 months
  Change in Pulse rate(beats per min)
Respiratory rate(breaths per min) | 12 months
  Change in Respiratory rate(breaths per min)
temperature(℃) | 12 months
  Change in temperature(℃)
EKG | 12 months
  EKG result(normal or abnormal)

OTHER OUTCOMES:
Change from the baseline in the total score of PSP-rating scale | 18 months
  Change from the baseline in the total score of PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 72 weeks (18 months) of investigational product administration. The possible total scores range from 0 to 100 with a higher score indicating severely impaired cognitive function.
Change from the baseline in the score of each domain of the PSP-rating scale | 18 months
  Change from the baseline in the score of each domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 72 weeks (18 months) and 24 weeks (6 months) of investigational product administration. Each domain is rated from different range (0 to 8, 16, 20 or 24) with a higher total score indicating severely impaired cognitive function.
Change from the baseline in the score of each item of the PSP-rating scale | 18 months
  Change from the baseline in the score of each item of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 72 weeks (18 months) of investigational product administration. Each item is rated from different range (0 to 2 or 4) with a higher total score indicating severely impaired cognitive function.
Change from the baseline in the Montreal Cognitive Assessment - Korea (MoCAK) | 18 months
  Change from the baseline in the Montreal Cognitive Assessment - Korea (MoCAK) after 72 weeks (18 months) of investigational product administration. The possible total scores range from 0 to 30 with a higher score indicating greater cognitive function.
Change from the baseline in the Korean Frontal Assessment Battery (K-FAB) | 18 months
  Change from the baseline in the Korean Frontal Assessment Battery (K-FAB) after 72 weeks (18 months) of investigational product administration. The possible total scores range from 0 to 18 with a higher score indicating greater cognitive function.
Change from the baseline in the England & Schwab Activity of Daily Living (ES ADL) scale | 18 months
  Change from the baseline in the England & Schwab Activity of Daily Living (ES ADL) scale after 72 weeks (18 months) of investigational product administration. The possible total scores range from 0 (complete dependence) to 100% (complete independence) based on the level of independence.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Jae Kim, Study Chair — GemVax & Kael
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No